CLINICAL TRIAL: NCT04769102
Title: Effect of Different Seat Cushions Adaptation on Upper Extremity Function in Children With Spastic Cerebral Palsy
Brief Title: Seat Cushions Adaptations on Upper Extremity Function In Cerebral Palsy Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hamada Ahmed, lecture of physical therapy, Biomechanic department, Faculty of Physical Therapy , Cairo Uni, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003018
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy
Keywords: seat cushions, upper extremity , cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spastic Cerebral Palsy (Experimental): spastic Cerebral palsy children will be adapted in adaptive seat with flat and then Contoured cushions while kinematic changes of upper limb reaching movement are monitored through video capture with kinovea 2D software motion analysis system.
  Interventions: Device: seat cushions

INTERVENTIONS:
Device: seat cushions — flat versus contoured customized seat cushions

SUMMARY:
As the seating adaptations, ranging from simple to complex, standard and customized may facilitate optimal health and maximize functional participation despite limited postural control; the study will be conducted for determine the effect of contoured cushions as a seat adaptation on upper extremity function in children with spastic cerebral palsy and compare between the effect of flat cushion and contoured cushion in adaptive seating system on upper extremity function in children with spastic cerebral palsy.

DETAILED DESCRIPTION:
As research continues to reveal the efficacy of ramped and contoured cushions on postural stability and alignment (Macdonald et al.,2015), it is likely that it will become accepted that such modifications will affect the UL functional level , mobility and rang of motion. Therefore, the purpose of this study was to examine the effect of contoured cushions as adaptive seating intervention on Upper extremity function in children with spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

1. Their age ranged from three to six years old .
2. Spasticity ranged from 1+ to 2 grade according to Modified Ashwarth Scale .
3. All children should be able to sit on the adaptive seat while head is upright independently and hands are free; preliminary test by Gross Motor Functional Measurement (GMFM) scale ranged score from ( 21 to 25 ) in sitting domain.

Exclusion Criteria:

Any child with the following criteria will be directly excluded from the evaluation for the consistency of the sample and statistically obtained results:

1. Visual and/or auditory defects which interfere with upper extremity functions.
2. Fixed deformity of one or both upper limbs which limit passive ROM in shoulder and elbow.
3. Children with mixed type, dyskinetic or ataxic cerebral palsy are excluded.
4. surgical intervention in both upper limbs or botulinum toxin injection in the last 6 months before the time of assessment .
5. Any recent trauma of one or Both upper limbs.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Angular kinematic changes in Upper extremity rang of motion in parallel to functional changes will be addressed while seat adaptations( flat and contoured cushions) will be applied for same participant. | within 30 to 60 minutes
  angular kinematic changes ( by degrees) will be measured by kinovea 2D software

CONTACTS AND LOCATIONS:
Overall Officials: Faten H. Abd El Azeem, Phd, Study Director — proffesor of peadiatric physical therapy Cairo Uni
Locations (1):
- Out Patient Clinic of Faculty of Physical Therapy Cairo Uni, Cairo, Giza- Beenelsarayat, Egypt

IPD SHARING:
Plan to Share IPD: No